CLINICAL TRIAL: NCT02685449
Title: Insulin Requirement for Pure- Protein Meal in Children With Type 1 Diabetes Treated With Continuous Subcutaneous Insulin Infusion - a Cross-over, Randomized Trial.
Brief Title: Insulin Requirement for Pure-protein Meal in Children With Type 1 Diabetes on Insulin Pumps.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Białko_5h
Record Dates: First submitted 2016-02-12; First posted 2016-02-18 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes type1
Keywords: diabetes type 1; insulin pump; prandial insulin requirement; pure protein meal; high protein meal; square bolus; square-wave bolus; insulin bolus; dietary protein
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin glulisine; Insulin Aspart; Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A (Placebo Comparator): On the first study day, insulin bolus was not given before a standardized pure protein meal. On the second day, pre-breakfast insulin was given as a square-wave bolus before the same standardized pure protein meal.
  The fat-protein-insulin ratio on both study days were identical to the patient's ratio when entering trial.
  Kind of study bolus insulin will be a rapid-acting insulin analog same as previously used by the participant (before entering the trial) - insulin aspart, insulin lispro or insulin glulisine
  Interventions: Drug: Insulin glulisine; Drug: Insulin aspart; Drug: Insulin lispro
- group B (Active Comparator): On the first study day, pre-breakfast insulin was given as a square-wave bolus before a standardized pure protein meal. On the second day, insulin bolus was not given before the same standardized pure protein meal.
  The fat-protein-insulin ratio on both study days were identical to the patient's ratio when entering trial.
  Kind of study bolus insulin will be a rapid-acting insulin analog same as previously used by the participant (before entering the trial) - insulin aspart, insulin lispro or insulin glulisine
  Interventions: Drug: Insulin glulisine; Drug: Insulin aspart; Drug: Insulin lispro

INTERVENTIONS:
Drug: Insulin glulisine — A kind of study bolus insulin will be insulin aspart if participant used insulin aspart before entering the trial
  Other Names: Apidra®
Drug: Insulin aspart — A kind of study bolus insulin will be insulin lispro if participant used insulin lispro before entering the trial
  Other Names: NovoRapid®
Drug: Insulin lispro — A kind of study bolus insulin will be insulin lispro if participant used insulin lispro before entering the trial
  Other Names: Humalog®

SUMMARY:
This is a randomized, cross-over study. The aim of this study is to compare the post-prandial glycaemic variability after pure protein meal following with an administration of square-wave bolus of meal-insulin or without any meal-insulin bolus on the other day.

Prolonged post-prandial glycaemic variability will be identified using the self-monitoring of blood glucose (10-point curve) and CGMS.

DETAILED DESCRIPTION:
The square-wave bolus (for meals rich in fat and/or protein) is evenly delivered over several hours as programmed by the patient. The required insulin dose will be calculated based on patient's insulin-exchange ratio. Pure protein meal will be given 3 hours after a first breakfast.

To provide the minimal impact of the previous breakfast, all patients will receive up to 120 kcal of carbohydrates and <100 kcal from protein and fat for the first breakfast (without any extended bolus) Patients receive a standardized pure protein meal at a second breakfast time. Meal insulin will be given as a square bolus or no meal -insulin will be given at all. The 5h post-meal glucose excursions will be recorded by self-blood glucose measurements (SMBG) (every 30 minutes) and continuous glucose monitoring system (CGMS). The intervention is taking part under in-patient clinical conditions.

ELIGIBILITY:
Inclusion Criteria:

* duration of type 1 diabetes longer than 12 months
* insulin pump therapy longer than 3 months
* written informed consent by patients and parents
* insulin requirement more than 0,5 units/kg/day

Exclusion Criteria:

* diabetes related complications (e.g. nephropathy)
* chronic kidney diseases
* any disease judged by the investigator to affect the trial
* withdrawal of consent to participate in the study

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Postprandial glycemia | 30 minutes after the meal
  Post-prandial blood glucose excursions measured by self monitoring of blood glucose (SMBG)
Postprandial glycemia | 60 minutes after the meal
  Post-prandial blood glucose excursions measured by self monitoring of blood glucose (SMBG)
Postprandial glycemia | 90 minutes after the meal
  Post-prandial blood glucose excursions measured by self monitoring of blood glucose (SMBG)
Postprandial glycemia | 120 minutes after the meal
  Post-prandial blood glucose excursions measured by self monitoring of blood glucose (SMBG)
Postprandial glycemia | 150 minutes after the meal
  Post-prandial blood glucose excursions measured by self monitoring of blood glucose (SMBG)
Postprandial glycemia | 180 minutes after the meal
  Post-prandial blood glucose excursions measured by self monitoring of blood glucose (SMBG)
Postprandial glycemia | 210 minutes after the meal
  Post-prandial blood glucose excursions measured by self monitoring of blood glucose (SMBG)
Postprandial glycemia | 240 minutes after the meal
  Post-prandial blood glucose excursions measured by self monitoring of blood glucose (SMBG)
Postprandial glycemia | 270 minutes after the meal
  Post-prandial blood glucose excursions measured by self monitoring of blood glucose (SMBG)
Postprandial glycemia | 300 minutes after the meal
  Post-prandial blood glucose excursions measured by self monitoring of blood glucose (SMBG)

SECONDARY OUTCOMES:
Hypoglycemia episodes | 5-hour study period
  Hypoglycemia defined as a plasma glucose concentration below 65 mg/dl with or without symptoms
Glucose Area Under the Curve (AUC) | 5-hour study period
  Measurements based on CGMS
Mean amplitude of glycemic excursion | 5-hour study period
  measurements based on SMBG
The difference between the maximum and baseline glucose level | 5-hour study period
  Post-prandial blood glucose excursions measured by self monitoring of blood glucose (SMBG)

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Dżygało, Principal Investigator — Department of Pediatrics, Warsaw Medical University; Kamila Indulska, Study Director — University of Alberta; Agnieszka Szypowska, Study Chair — University of Alberta
Locations (1):
- Medical University, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No